CLINICAL TRIAL: NCT01391741
Title: The Effect of High-Volume Walking With Visual Cues on Gait in People With Parkinson´s Disease. A Randomized Controlled Trial
Brief Title: The Effect of High-Volume Walking With Visual Cues (VC) in Parkinson´s Disease (PD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Iceland (Other)
Collaborators: The Icelandic Parkinson´s Association. (Other); Icelandic Physiotherapy Association (Other)
Responsible Party: Andri Thor Sigurgeirsson/Mr., University of Iceland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 123SmOkE
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2010-03

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s Disease; Walking; Exercise; Automaticity; Dual Task; Visual Cues; Cueing; Neuroplasticity; Gait analysis
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walking with visual cues (Experimental): Walking with visual cues for 30 minutes, 4 times a week for 4 weeks
  Interventions: Other: Visual Cues
- Walking without visual cues (Active Comparator): Walking without visual cues, but verbal encouragement twice a week to take longer steps, for 30 minutes, 4 times a week for 4 weeks.
  Interventions: Other: Walking without visual cues

INTERVENTIONS:
Other: Visual Cues — Walking with visual cues for 30 minutes, 4 times a week for 4 weeks
  Arms: Walking with visual cues
Other: Walking without visual cues — Walking without visual cues, but verbal encouragement twice a week to take longer steps, for 30 minutes, 4
  Arms: Walking without visual cues

SUMMARY:
People with disease (PD) tend to walk with short steps, decreased velocity, and increased stride time variability. Short steps and increased variability are related to greater fall risk. In addition, concurrent performance of a cognitive task (dual-task (DT)) has marked effects on gait in people with PD which is considered to reflect an impaired automaticity of gait.

Objective: To investigate short and long term effects of high-volume walking with visual spatial cues (VSC) on gait variables, automaticity, and functional mobility, in people with Parkinson´s Disease (PD), compared with walking without VSC.

ELIGIBILITY:
Inclusion Criteria:

* a confirmed diagnosis of PD according to the UK Parkinson´s Disease Society Brain Bank Clinical Diagnostic Criteria (18)
* <80 years of age
* community residing
* Hoehn and Yahr (HY) stage 2-3
* Mini Mental State Examination (MMSE) score of >23
* ability to walk without walking aids for a total of 20 minutes over a 30-minute period

Exclusion Criteria:

* major modifications of Parkinson´s medication (Madopar >200 mg/d or >20% increase in Dopamine agonists) 3 weeks prior to baseline assessment
* comorbidities or disabilities, which might influence walking
* a history of brain surgery

Max Age: 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Change in Step Length | Before, after and 3 months after a 4 week training period
Change in Gait Velocity | Before, after and 3 months after a 4 week training period
Change in Stride Time Variability | Before, after and 3 months after a 4 week training period

SECONDARY OUTCOMES:
Change in Timed Up & Go (seconds) | Before, after and 3 months after a 4 week training period

CONTACTS AND LOCATIONS:
Overall Officials: Andri T Sigurgeirsson, M.Sc., Principal Investigator — University of Iceland / Reykjalundur Rehabilitation Center
Locations (1):
- Reykjalundur Rehabilitation Center, Mosfellsbaer, Iceland